CLINICAL TRIAL: NCT05203419
Title: A Two-part, Randomized, Investigator- and Participant- Blinded, Placebo-controlled, Multiple Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MHS552 in Adult Participants With Systemic Lupus Erythematosus (SLE)
Brief Title: Multiple Ascending Dose Study of MHS552 in Adults Participants With Systemic Lupus Erythematosus (SLE)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMHS552D12101; 2021-003520-33 (EudraCT Number)
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Systemic Lupus Erythematosus, Lupus, autoimmune disease, inflammatory disease, inflammation
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Part A: Cohort 1 - MHS552 low dose (Experimental): Participants will receive MHS552 low dose once weekly subcutaneously for 4 weeks
  Interventions: Drug: MHS552
- Part A: Cohort 1, 2, 3 - Placebo (Placebo Comparator): Participants will receive placebo once weekly subcutaneously for 4 weeks
  Interventions: Drug: Placebo
- Part A: Cohort 2 - MHS552 medium dose (Experimental): Participants will receive MHS552 medium dose once weekly subcutaneously for 4 weeks
  Interventions: Drug: MHS552
- Part A: Cohort 3 - MHS552 high dose (Experimental): Participants will receive MHS552 high dose once weekly subcutaneously for 4 weeks
  Interventions: Drug: MHS552
- Part B: MHS552 (Experimental): Participants will receive MHS552 (dose to be determined) once weekly subcutaneously for 12 weeks
  Interventions: Drug: MHS552
- Part B: Placebo (Placebo Comparator): Participants will receive placebo once weekly subcutaneously for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MHS552 — MHS552 will be administered once weekly as subcutaneous injection for 4 weeks (Part A) or 12 weeks (Part B)
  Arms: Part A: Cohort 1 - MHS552 low dose; Part A: Cohort 2 - MHS552 medium dose; Part A: Cohort 3 - MHS552 high dose; Part B: MHS552
Drug: Placebo — Placebo will be administered once weekly as subcutaneous injection for 4 weeks (Part A) or 12 weeks (Part B)
  Arms: Part A: Cohort 1, 2, 3 - Placebo; Part B: Placebo

SUMMARY:
The purpose of this two-part multiple ascending dose study is to evaluate the safety and tolerability of multiple doses of MHS552 in adults with mild to moderately active Systemic Lupus Erythematosus (SLE). Participants will be treated for 4 or 12 weeks followed by an 8-week follow-up period.

DETAILED DESCRIPTION:
This was a Phase 1b, randomized, placebo-controlled, participant- and investigator- blinded, two-part non-confirmatory multiple ascending dose (MAD) study in adult patients aged 18-65 (inclusive) with active SLE disease (mild-moderate).This MAD study was planned to be conducted in two parts, Part A and Part B sequentially, but the study was terminated before Part B was initiated.

In Part A, after a screening period of up to 6 weeks, participants were randomized (in a 3:1 ratio) to MHS552 or placebo administered subcutaneously (s.c.) weekly for four weeks of treatment. Part A was planned to consist of up to 3 cohorts (low, medium, high dose). Due to termination of the trial, Part A consisted of 2 cohorts (low and medium doses). Participants were followed-up during 8 weeks post last dose. The total duration of study participation of Part A was approximately 120 Days.

In Part B (not started due to termination of the trial), it was planned that after a screening period of up to 28 days, approximately 12 participants to be randomized (in a 2:1 ratio) to MHS552 or placebo administered s.c. weekly for 12 weeks of treatment (dose to be confirmed).

ELIGIBILITY:
Inclusion Criteria:

* Fulfills the 2019 EULAR/American College of Rheumatology (ACR) classification criteria for SLE at least 3 months prior to and at screening.
* Patients with mild or moderately active SLE (SLEDAI-2K between 3 and 10, inclusive) at screening. Patients with cutaneous lupus are eligible as long as they satisfy the criteria for systemic lupus.
* Patients must be on stable dose(s) of at least one of the following medications, unless the medication has been discontinued due to intolerance, inadequate response, or patient/physician decision:

  * steroid at a dose ≥ 5mg but <30 mg of prednisone (or equivalent) per day,
  * antimalarial (hydroxychloroquine/chloroquine/quinacrine) or thalidomide,
  * disease modifying anti-rheumatic drugs (DMARDs):
  * methotrexate (MTX),
  * azathioprine (AZA),
  * mizoribine,
  * mycophenolate derivates. Steroid dose must be stable for at least 4 weeks prior to the first dosing. The dose of the other medications above must be stable for at least 12 weeks prior to the first dosing. If the patient is not on any medications listed above, they must have been off these medications for at least 12 weeks prior to dosing.

Exclusion Criteria:

* History of hypersensitivity to drugs of similar biological class, IL-2 protein analogues, or hypersensitivity to any components of the study drug, or history of severe hypersensitivity reaction or anaphylaxis to biological agents, e.g. human monoclonal antibody.
* Patients with central nervous system (CNS) lupus, active Lupus Nephritis, any type of lupus flare requiring pulse steroid or immunosuppressive therapy with cyclophosphamide, rituximab, calcineurin inhibitors, or others except those permitted in the inclusion criteria.
* Systemic autoimmune disease other than lupus, which would interfere with participation in the study according to the Investigator's judgement. Treated, stable Hashimoto's thyroiditis is not exclusionary.
* Any of the following abnormal laboratory values at Screening or pre-dose Day 1 assessment:

Hemoglobin levels below 8.0 g/dL at screening Eosinophil count >700 mm3 or >2 X Upper Limit of Normal (ULN), whichever is lower.

- History of capillary leak syndrome (CLS).

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-06-04 (Actual); Study Completion 2023-06-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse events (AEs) and Serious Adverse events (SAEs) | Part A: up to 12 weeks; Part B: up to 20 weeks
  Numbers of participants with AEs and SAEs, and other safety data such as vital signs, electrocardiograms (ECG) and laboratory results

SECONDARY OUTCOMES:
Area Under Plasma Concentration-time Curve calculated to the end of a dosing interval (AUCtau) for MHS552 | Part A: up to Day 78; Part B: up to Day 134
  Characterize the AUCtau profile following multiple doses of MHS552
Maximum Observed Blood Concentrations (Cmax) for MHS552 | Part A: up to Day 78; Part B: up to Day 134
  Characterize the Cmax profile following multiple doses of MHS552
Time to Reach Maximum Blood Concentrations (Tmax) of MHS552 | Part A: up to Day 78; Part B: up to Day 134
  Characterize the Tmax profile profile following multiple doses of MHS552

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18163
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2084